CLINICAL TRIAL: NCT00465465
Title: A Dose Selection Study Evaluating the Safety and Immunogenicity of 2 Different Doses of a New TB Vaccine, MVA85A, in Healthy Volunteers Who Have Previously Been Vaccinated With BCG
Brief Title: A Study of 2 Doses of a New TB Vaccine, MVA85A, in Healthy Volunteers Previously Vaccinated With BCG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Dr Helen McShane, University of Oxford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB009
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2008-03

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; TB; MVA 85A; BCG
MeSH Terms: conditions — Tuberculosis | interventions — MVA 85A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Dose of 1 x 10^7
  Interventions: Biological: MVA 85A
- 2 (Active Comparator): Dose of 1 x 10^8
  Interventions: Biological: MVA 85A

INTERVENTIONS:
Biological: MVA 85A — i.d. injection

SUMMARY:
The dose of recombinant MVA used in the TB trials to date is relatively low compared with other trials using recombinant MVAs which have used up to 2.5 x 108pfu (A Hill, personal communication). Having demonstrated safety and immunogenicity of 5 x 107pfu of MVA85A, we now need to perform a dose optimization study, prior to commencing larger scale Phase II and III studies in South Africa. We will vaccinate 12 volunteers with a dose half a log lower than the dose we are currently using, i.e. 107pfu MVA85A, and 12 volunteers with a dose half a log higher, i.e. 108pfu.

DETAILED DESCRIPTION:
MVA85A (at a dose of 5 x 107pfu) has been administered to 41 healthy volunteers in the UK and 17 healthy volunteers in The Gambia, with no serious adverse events. We have designed our Phase I studies to allow for a vaccination of volunteer groups sequentially with a step-wise increase in mycobacterial exposure, in order to minimize the possibility of a Koch reaction. A Koch reaction describes the development of immunopathology in a person or animal with tuberculosis, when an exaggerated immune response to M.tb is stimulated. It was described in patients with TB disease when Koch performed his original studies employing mycobacteria as a type of therapeutic vaccination. It has now been demonstrated in the mouse model of therapeutic vaccination (Taylor, 2003). Available animal data suggest that these reactions do not occur in mice latently infected with M.tb, suggesting that such reactions may correlate with high bacterial load and that the Koch phenomenon may not pose a problem for vaccination of healthy albeit latently infected humans. We started these studies in healthy volunteers who were as mycobacterially naïve as possible. They were skin test negative and Elispot negative for PPD, ESAT 6 and CFP10, and had not had previously been vaccinated with BCG. We have now completed studies in the UK vaccinating volunteers previously vaccinated with BCG (McShane, 2004). These volunteers are excluded if their Mantoux test is greater than 15 millimeters. These studies are ongoing in The Gambia. The group we are currently recruiting for on this increasing mycobacterial spectrum are healthy volunteers who are latently infected with M.tb.

Decision matrix for selecting MVA85A dose

1. If reducing the dose of MVA85A results in reduced immunogenicity, we could use either the 5x107 or 108 dose, and would select the lower of these on the grounds of safety.
2. If increasing the dose of MVA85A increases the incidence of side-effects, we could use either the 5x107 or 107 dose, and we would use the higher of these on the grounds of immunogenicity.
3. If increasing the dose of MVA85A results in increased immunogenicity and no increase in side-effects, we could use either the 5x107 or 108 dose in subsequent trials
4. If reducing the dose of MVA85A results in no reduction in immunogenicity we could use either the 107 or 5x107 dose in subsequent trials
5. If all three doses are equally safe and immunogenic we will use either the low or 5x107 dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Resident in or near Oxford for the duration of the vaccination study
* Willingness to allow the investigators to discuss the volunteer's medical history with the volunteer's GP
* Screening Elispot negative (less than 10 sfc/million PBMC) for all 3 ESAT6 peptide pools and all 3 CFP10 peptide pools
* Mantoux test not greater than 15 millimetres
* For females only, willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day of vaccination
* Agreement to refrain from blood donation during the course of the study
* Written informed consent
* Willingness to undergo an HIV test

Exclusion Criteria:

* Any deviation from the normal range in biochemistry or haematology blood tests or in urine analysis as defined in Appendix I
* Mantoux greater than 15 millimetres
* Prior receipt of a recombinant MVA or Fowlpox vaccine
* Use of any investigational or non-registered drug, live vaccine or medical device other than the study vaccine within 30 days preceding dosing of study vaccine, or planned use during the study period
* Administration of chronic (defined as more than 14 days) immunosuppressive drugs or other immune modifying drugs within six months of vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection and asplenia
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* Evidence of cardiovascular disease
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of insulin requiring diabetes mellitus
* Chronic or active neurological disease requiring ongoing specialist supervision
* Chronic gastrointestinal disease requiring ongoing specialist supervision
* History of > 2 hospitalisations for invasive bacterial infections (pneumonia, meningitis)
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Evidence of serious psychiatric condition
* Any other on-going chronic illness requiring hospital specialist supervision
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Pregnant or lactating female
* Female who is willing or intends to become pregnant during the study
* Any history of anaphylaxis in reaction to vaccination
* Inability to give informed consent
* PI assessment of lack of willingness to participate and comply with all requirements of the protocol
* Any other finding which in the opinion of the investigator would significantly increase the risk of having an adverse outcome from participating in this protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To assess the safety and immunogenicity of 2 different doses of intradermal vaccination of MVA85A, 10^7pfu and 10^8pfu, when administered to healthy subjects who have previously been vaccinated with BCG | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, CCVTM, Churchill Hospital, Oxford, Oxfordshire, United Kingdom